CLINICAL TRIAL: NCT01828931
Title: Effectiveness of Intensive Lifestyle Interventions in the Management of Diabetes in Individuals With Psychosis
Brief Title: Lifestyle Intervention for Diabetes and Weight Management in Psychosis
Acronym: Healthy_LIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Principal Investigator, Margaret Hahn, Staff Psychiatrist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 151/2012
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes Mellitus; Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Bipolar I Disorder; Substance-induced Psychosis; Psychotic Disorders; Major Depressive Disorder
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Schizophrenia; Psychotic Disorders; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Standard care provided via participants' family physicians, diabetes nurses, and psychiatrists.
  Interventions: Other: Usual Care
- Lifestyle Intervention (Experimental): A lifestyle intervention based on the Look AHEAD study intervention, involving counselling related to dietary and physical activity habits.
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention — A lifestyle intervention (LI) aimed at reducing caloric intake and increasing physical activity
  Arms: Lifestyle Intervention
Other: Usual Care — Care as usual
  Arms: Usual Care

SUMMARY:
The rate of type-2 diabetes mellitus (T2DM) is at least 2-3 times higher in persons with psychotic illnesses than in the general population. Life expectancy of individuals with psychosis is also 20-25 years less than the general population, primarily due to premature onset of cardiovascular disease (CVD). Despite the high risk for T2DM and CVD, psychotic illness has been an exclusion criterion in all large-scale studies of diabetes prevention and management. We propose a 3-year randomized controlled trial examining the effectiveness of a lifestyle intervention (LI) aimed at reducing caloric intake and increasing physical activity in overweight or obese individuals (N=150) suffering from both a psychotic illness and T2DM. Weight and glycemic control will be the primary outcome variables. It is hypothesized that a significant weight reduction and improvement in glycemic control will be found in those who receive the LI relative to those who do not.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 70 years (inclusive)
2. DSM-IV-TR diagnosis of one of the psychotic disorders listed above
3. Body Mass Index (BMI) > 25 kg/m2 at the time of enrollment
4. Clearly documented diagnosis of type-2 diabetes mellitus or prediabetes
5. Ability to provide informed consent
6. No medical contraindication to participation in weight reduction / exercise program, determined in consultation with their primary care physician
7. Female participants, of childbearing potential, using a medically accepted means of contraception

Exclusion Criteria:

1. Inability to give informed consent
2. Currently enrolled in a formal structured weight management program
3. Currently being prescribed medication specifically for weight loss
4. Participants with unstable or active cardiovascular illnesses (myocardial infarction, CHF, etc), active or end-stage renal disease, unstable thyroid disease, etc.
5. Recurrent episodes of diabetic ketoacidosis, seizure or coma without warning or severe hypoglycemia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-12; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Weight | 52 weeks
HbA1c levels | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Margaret K Hahn, M.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided